CLINICAL TRIAL: NCT00018811
Title: Psychological Assessment and Treatment of Chronic Benign Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHBS-001-99S2
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2003-12

CONDITIONS: Headache; Migraine; Tension Headache; Stress Headache; Vascular Headache
Keywords: Relaxation Techniques; Behavior Therapy Feedback; Psychophysiology
MeSH Terms: conditions — Headache; Migraine Disorders; Tension-Type Headache; Vascular Headaches | interventions — Relaxation Therapy

INTERVENTIONS:
Behavioral: Relaxation training & thermal biofeedback
Behavioral: Surface EMG biofeedback

SUMMARY:
Subjects with chronic migraine or tension headaches will receive 12 sessions of biofeedback or relaxation training after fulfilling screening, intake interviews, & psychological testing requirements. They will chart headache pain, anger level, & medication usage throughout baseline, treatment, and 3 month follow-up periods.

Migraine sufferers will receive a combination of progressive muscle relaxation training and thermal biofeedback (learning to warm hands). Subjects are randomly assigned to receive treatment either in the office with the therapist or from another room (where communication will be over a computer). The research is designed to compare the effectiveness of treatment based on location.

Tension headache sufferers will receive training in how to reduce their muscle tension levels. They will be randomly assigned to have equipment monitor muscle tension levels either in the forehead or shoulder regions. The research is designed to compare the effectiveness of feedback to the forehead versus the shoulder muscles.

ELIGIBILITY:
Subjects must be at least 18 years old and have chronic headaches of any of the following types: migraine, coexisting migraine/tension, or tension. Participants must be intellectually intact and have no significant physical, neurological, or psychological problems. They must have seen a physician for their headaches within the past year. They must successfully complete screening/interview/testing process prior to admission to treatment.

All vascular headache subjects must meet the criteria for chronic migraine or coexisting migraine and tension type headache as set forth by the Headache Classification Committee of the International Headache Society.

All tension headache subjects must meet the criteria for either episodic or chronic tension headache set forth by the Headache Classification Committee, as well as the Ad Hoc Committee's criteria for tension headache.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veterans Affairs Medical Center, Augusta, Georgia, United States